CLINICAL TRIAL: NCT03313271
Title: China Lymphoma Patient Registry Study
Acronym: CLAP
Status: Recruiting | Type: Observational
Sponsor: Jun Zhu (Other)
Collaborators: Peking University First Hospital (Other); Tianjin Medical University Cancer Hospital (Unknown); Zhejiang Cancer Hospital (Other); Heilongjiang Cancer Hospital (Unknown); Sipai(Beijing)Network Technology Co Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Jun Zhu, Director of lymphoma department, Peking University
Organization: Peking University (Other)
Other Study IDs: h-yx-bj-16003
Record Dates: First submitted 2017-10-11; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma
Keywords: lymphoma; CLAP; China; patient registry
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- a cohort of patients with lymphoma in China: establish a cohort of patients with lymphoma in China and follow up the patients for a long period of time

SUMMARY:
Lymphoma is the most common hematologic tumor. It is derived from lymphoid tissue, including Hodgkin's lymphoma(HL) and non Hodgkin's lymphoma(NHL). The treatment of lymphoma includes chemotherapy, radiotherapy, stem cell transplantation, targeted therapy and surgery etc. With the progress of treatment, the survival rate of lymphoma patients has been improved. But the 5 year survival rate of lymphoma in China is shorter than that in United States. The reason is that there is still a gap between China and the United States in disease screening, diagnosis and treatment.

Observational studies, especially cohort studies, are important tools for understanding disease progression, treatment, and prognosis in the real world. Observational cohort studies which involve over 500 patients are currently launched by South Korea and the United States. China, which has more patients, doesn't have a cohort of patients with lymphoma. So the primary objective of this study was to establish an observational cohort of patients with lymphoma in China and follow up the patients for a long period of time to provide basic support for clinical research and drug development, and continuously improve patient outcomes and quality of life. The secondary objective is to collect information about diagnosis, treatment, follow-up and prognosis of lymphoma.

DETAILED DESCRIPTION:
Lymphoma is the most common hematologic tumor. It is derived from lymphoid tissue, including Hodgkin's lymphoma(HL) and non Hodgkin's lymphoma(NHL). The treatment of lymphoma includes chemotherapy, radiotherapy, stem cell transplantation, targeted therapy and surgery etc. With the progress of treatment, the survival rate of lymphoma patients has been improved. But the 5 year survival rate of lymphoma in China is shorter than that in United States. The reason is that there is still a gap between China and the United States in disease screening, diagnosis and treatment.

Observational studies, especially cohort studies, are important tools for understanding disease progression, treatment, and prognosis in the real world. Observational cohort studies which involve over 500 patients are currently launched by South Korea and the United States. China, which has more patients, doesn't have a cohort of patients with lymphoma. So the primary objective of this study was to establish an observational cohort of patients with lymphoma in China and follow up the patients for a long period of time to provide basic support for clinical research and drug development, and continuously improve patient outcomes and quality of life. The secondary objective is to collect information about diagnosis, treatment, follow-up and prognosis of lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* The disease was diagnosed by Hodgkin's or non Hodgkin's lymphoma
* 18 years of age or older at diagnosis
* The diagnosis was confirmed within 6 months before admission
* Informed consent was obtained

Exclusion Criteria:

* There are no special exclusion criteria in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma patients in 5 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Characteristics of lymphoma in China， | 5 years
  Understand the characteristics of lymphoma in China,such as the distribution of sex,age,histological type and clinical stage etc

SECONDARY OUTCOMES:
Overall survival | 10 years
  Overall survival is defined as the time from disease to death

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Ph D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Zeng H, Zheng R, Guo Y, Zhang S, Zou X, Wang N, Zhang L, Tang J, Chen J, Wei K, Huang S, Wang J, Yu L, Zhao D, Song G, Chen J, Shen Y, Yang X, Gu X, Jin F, Li Q, Li Y, Ge H, Zhu F, Dong J, Guo G, Wu M, Du L, Sun X, He Y, Coleman MP, Baade P, Chen W, Yu XQ. Cancer survival in China, 2003-2005: a population-based study. Int J Cancer. 2015 Apr 15;136(8):1921-30. doi: 10.1002/ijc.29227. Epub 2014 Oct 3. PMID 25242378
- [Background] De Angelis R, Sant M, Coleman MP, Francisci S, Baili P, Pierannunzio D, Trama A, Visser O, Brenner H, Ardanaz E, Bielska-Lasota M, Engholm G, Nennecke A, Siesling S, Berrino F, Capocaccia R; EUROCARE-5 Working Group. Cancer survival in Europe 1999-2007 by country and age: results of EUROCARE--5-a population-based study. Lancet Oncol. 2014 Jan;15(1):23-34. doi: 10.1016/S1470-2045(13)70546-1. Epub 2013 Dec 5. PMID 24314615
- [Background] Australian Institute of Health and Welfare. Cancer survival and prevalence in Australia: period estimates from 1982 to 2010. Asia Pac J Clin Oncol. 2013 Mar;9(1):29-39. doi: 10.1111/ajco.12062. PMID 23418847